CLINICAL TRIAL: NCT02531321
Title: Effects of Protease Inhibitor Use on Combined Oral Contraceptive Pharmacokinetics and Pharmacodynamics in HIV-positive Women
Brief Title: Protease Inhibitors and Combined Oral Contraceptive Pharmacokinetics and Pharmacodynamics
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Nicole Bender, Assistant Professor, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-15-00112
Record Dates: First submitted 2015-08-19; First posted 2015-08-24 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Contraception; HIV
MeSH Terms: interventions — ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ritonavir (Experimental): Participants taking antiretroviral regimens including ritonavir-boosted protease inhibitors will take a combined oral contraceptive containing 150mcg levonorgestrel and 30mcg ethinyl estradiol for 21 days.
  Interventions: Drug: Levonorgestrel and Ethinyl Estradiol
- Control (Active Comparator): Participants taking antiretroviral regimens known not to interact with oral contraceptives will take a combined oral contraceptive containing 150mcg levonorgestrel and 30mcg ethinyl estradiol for 21 days.
  Interventions: Drug: Levonorgestrel and Ethinyl Estradiol

INTERVENTIONS:
Drug: Levonorgestrel and Ethinyl Estradiol — All participants will take a combined oral contraceptive containing 150mcg levonorgestrel and 30mcg ethinyl estradiol for 21 days. Pharmacokinetics and pharmacodynamics will be compared between participants using antiretroviral regimens including ritonavir-boosted protease inhibitors and those using regimens that do not interact with oral contraceptives.

SUMMARY:
The project is a two-arm prospective cohort and pharmacokinetic study comparing levonorgestrel and ethinyl estradiol pharmacokinetics in HIV-positive women taking antiretroviral regimens that include ritonavir to those in women who take regimens known not to interact with combined oral contraceptives. In addition, the prevalence of ovulation will be measured in each group. Participants will take a combined oral contraceptive containing levonorgestrel and ethinyl estradiol for 21 days, during which they will undergo twice-weekly serum progesterones. On the final day, they will complete a pharmacokinetic study. The investigators hypothesize that levonorgestrel levels, as measured by area-under-the-curve from 0 to 72 hours, will be increased in women on ritonavir, while ethinyl estradiol levels will be decreased and ovulation, defined by a serum progesterone of at least 3 ng/mL, will be unchanged.

This study will be the first to evaluate the effects of ritonavir on the pharmacokinetics of a combined oral contraceptive containing the progestin levonorgestrel. In addition, no previous studies have rigorously assessed ovulation in women taking protease inhibitors and combined oral contraceptives. As a result, this study will provide new information correlating pharmacokinetic changes with effects on ovulation.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Female
* Age 18-45
* Using any of the following medication regimens: no ARV medication, entry inhibitors, nucleoside reverse transcriptase inhibitors (NRTIs), integrase inhibitors, and CCR5 agonists. Acceptable NRTI combinations include zidovudine (ZDV), lamivudine (3TC), emtricitabine (FTC), didanosine (ddl), stavudine (d4T), abacavir (ABC), and tenofovir disoproxil fumarate (TDF)
* Ovulatory (mid-luteal progesterone >3ng/dL)
* Not planning to conceive during the study period
* Willing to abstain from grapefruit products
* If taking ritonavir, willing to use alternate non-hormonal contraception
* BMI < or = 40
* Able to consent in English or Spanish
* No change in medication regimen for at least 21 days prior to study entry and no planned change during the study period
* CD4 > or =200, and/or not considered profoundly immuncompromised by primary HIV provider

Exclusion Criteria:

* Using on the combination of ZDV at d4T
* Platelets <50,000
* AST or ALT > twice upper limit of normal
* Bilirubin > twice upper limit of normal
* Use of other CYP3A4 inducing or inhibiting medications
* Pregnant or breastfeeding in last 30 days
* Use of DepoProvera in last 180 days
* Use of any other hormonal contraception in last 30 days
* Undiagnosed vaginal bleeding or invasive cancer of the reproductive tract

  ->50% change in tobacco use in the last month
* Initiation or titration of methadone therapy in the last month
* Uncontrolled thyroid disease
* Contraindication to estrogen use
* Inability to comply with study protocol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ritonavir | Control
Started | 7 | 10
Completed | 5 | 10
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ritonavir | Control | Total
Number analyzed (Participants) | 5 | 10 | 15
Age, Continuous [Median (Full Range); unit: years] | 38 [29 to 41] | 34.5 [30 to 42] | 35 [29 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Levonorgestrel Area Under the Curve
Description: Levonorgestrel AUC from 0 to 72 hours
Time Frame: 24 days
Measure: Mean (Standard Deviation); unit: ng/mL*h
Arm/Group | Ritonavir | Control
Number analyzed (Participants) | 5 | 10
ng/mL*h | 321 (61) | 243 (83)
Statistical Analysis 1: Comparison: Ritonavir vs Control; Test type: Other — Unpaired t test with Welch's correction; p < .05, t-test, 2 sided

2. Secondary Outcome: Ethinyl Estradiol Area Under the Curve
Description: Ethinyl estradiol area under the curve from 0 to 72 hours
Time Frame: 24 days
Measure: Mean (Standard Deviation); unit: ng/mL*h
Arm/Group | Ritonavir | Control
Number analyzed (Participants) | 5 | 10
ng/mL*h | 3867 (976) | 3270 (744)

3. Secondary Outcome: Serum Progesterone Level >3ng/dL Reflecting Ovulation
Description: Progesterone >3ng/dL at any time during pill use
Time Frame: 21 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ritonavir | Control
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 0/7 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No